CLINICAL TRIAL: NCT07340307
Title: Application of Wrist-Ankle Acupuncture in Patients With Different Types of Pain Following Perianal Surgery: A Prospective Cohort Study
Brief Title: Application Effects of Wrist-Ankle Acupuncture in Patients With Different Types of Pain Following Perianal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHPutianU-015
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Wrist-Ankle Acupuncture
Keywords: Wrist-Ankle Acupuncture; Analgesia; Pain Management; Perianal abscess; hemorrhoids; anal fistula
MeSH Terms: conditions — Agnosia; Hemorrhoids; Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spastic pain group (Experimental): The pain in this group of patients was characterized as sphincter spasm pain. Postoperatively, patients received routine care and were administered wrist-ankle acupuncture when their pain score (VRS) reached ≥4 points (performed at standardized zones 1 and 6 of both lower limbs, once daily, with treatment duration adjusted based on symptom response). If the pain score (VAS) remained ≥4 points 30 minutes after treatment, analgesic medication was additionally administered.
  Interventions: Device: wrist-ankle acupuncture
- Acute incisional pain group (Experimental): The pain in this group of patients was characterized as acute incisional pain. Postoperatively, patients received routine care and were administered wrist-ankle acupuncture when their pain score (VRS) reached ≥4 points. The procedure was performed at standardized zones 1 and 6 of both lower limbs, once daily, with the treatment duration adjusted according to symptom response. If the pain score (VAS) remained ≥4 points 30 minutes after treatment, analgesic medication was additionally administered.
  Interventions: Device: wrist-ankle acupuncture

INTERVENTIONS:
Device: wrist-ankle acupuncture — Patients received routine postoperative care, including intravenous infusion of flurbiprofen (50 mg, twice daily), herbal sitz baths, and pain management education. When a patient's Verbal Rating Scale (VRS) score reached ≥4 points, Wrist-Ankle Acupuncture therapy was administered. The procedure involved superficial subcutaneous insertion of disposable sterile needles (0.25 mm × 25 mm) at zones 1 and 6 of both lower limbs. The needle body was inserted subcutaneously, leaving approximately 1-2 mm exposed externally, with the aim of avoiding the induction of soreness, numbness, distension, or pain. Needles were retained for 0.5-1 hour, with treatment administered once daily. The treatment course was adjusted based on the degree of symptom relief. If the Visual Analog Scale (VAS) score remained ≥4 points 30 minutes after initiating Wrist-Ankle Acupuncture treatment, analgesic medication was administered as prescribed.

SUMMARY:
This study is a prospective clinical observation designed to evaluate the analgesic effect of wrist-ankle acupuncture in patients with different types of pain after perianal surgery, as well as its applicability. A total of 60 eligible postoperative patients were enrolled, with inclusion criteria including age 18-75 years, postoperative Visual Analog Scale (VAS) score ≥4, clear consciousness, and signed informed consent. Exclusion criteria included pregnancy, history of needle fainting, skin lesions at the wrist or ankle, severe systemic diseases, inability to cooperate with follow-up, or participation in other clinical trials. Patients were divided into two groups according to the nature of pain: Group A (sphincter spasm pain, n=30) and Group B (acute incisional pain, n=30). All patients received routine postoperative care (including intravenous flurbiprofen infusion, traditional Chinese medicine soaking, and pain education), and wrist-ankle acupuncture was administered when pain intensity (Verbal Rating Scale, VRS) reached ≥4. The acupuncture method involved superficial subcutaneous insertion in zones 1 and 6 of both lower limbs using disposable sterile needles (0.25 mm × 25 mm). Needles were retained for 0.5-1 hour, once daily, with the treatment course adjusted based on symptom relief. If the VAS score remained ≥4 at 30 minutes post-treatment, adjunctive analgesic medication was administered as prescribed. Observation indicators included postoperative VRS scores, reduction in VAS scores at 5 and 30 minutes after wrist-ankle acupuncture treatment, frequency of analgesic medication use within the first 3 postoperative days, and the Clinical Postoperative Urinary Retention (POUR) score at 24 hours post-surgery. By comparing data between the two groups, the analgesic effect of wrist-ankle acupuncture was analyzed, and the influence of postoperative pain on the occurrence of urinary retention was explored.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years;
* Patients who underwent perianal surgery;
* Visual Analog Scale (VAS) score ≥4;
* Clear consciousness with the ability to articulate their sensations;
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Pregnant or lactating patients;
* Patients with a history of needle fainting or needle phobia;
* Patients with incomplete skin integrity at the wrist or ankle;
* Patients with comorbid systemic diseases, such as cardiac insufficiency or coagulation disorders;
* Patients unable to cooperate with follow-up;
* Patients currently participating in other clinical trials that may influence the outcomes of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | During the hospitalization period
  Pain assessment was conducted using the Visual Analog Scale (VAS). A 10-cm horizontal line was drawn on paper, with one end marked as "0" indicating "no pain" and the opposite end marked as "10" indicating "severe pain." The intermediate sections represented varying degrees of pain intensity. Patients were instructed to mark a point on the line based on their subjective perception of pain. Assessments were performed at 24 hours postoperatively, as well as at 5 minutes and 30 minutes after the administration of wrist-ankle acupuncture therapy. The reduction in Visual Analogue Scale（VAS） scores was recorded accordingly.

SECONDARY OUTCOMES:
Analgesic Medication Frequency | During the hospitalization period
  The frequency of use of postoperative analgesic medications, such as flurbiprofen, was recorded.
Clinical Postoperative Urinary Retention (POUR) Score | 7days postoperativelyacupuncture administration.
  The Clinical Postoperative Urinary Retention (POUR) scores of patients were observed and recorded at 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, China

IPD SHARING:
Plan to Share IPD: No
Based on a strict commitment to participant privacy protection, compliance with the terms of the ethical review protocol, and adherence to the sponsoring institution's policies, IPD from this study will not be shared at this time.